CLINICAL TRIAL: NCT07048041
Title: Comparison of Patient-Reported Outcomes and Functional Tests After Hip Replacement Surgery
Brief Title: Patient Scores and Functional Tests After Hip Surgery
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Elif AYGUN POLAT, Principal Investigator, Ordu University
Other Study IDs: ODU-SBFTR-AYGUNPOLAT-006
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Total Hip Replacement; Patient-Reported Outcomes
Keywords: Total Hip Arthroplasty; Patient-Reported Outcomes; Physical Performance Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total Hip Arthroplasty (THA) patients: Patients who underwent primary unilateral total hip arthroplasty at least 6 months prior and met all inclusion criteria. Participants were evaluated using patient-reported outcome measures and performance-based physical tests in a single session.
  Interventions: Other: Functional Assessment Battery

INTERVENTIONS:
Other: Functional Assessment Battery — Participants completed a series of validated patient-reported outcome questionnaires (Oxford Hip Score, WOMAC, SF-12) and physical performance tests (Timed Up and Go, Four Square Step Test, 4-Meter Gait Speed Test) during a single outpatient assessment session. No therapeutic or invasive interventions were performed.
  Other Names: Timed Up and Go; Four Square Step Test; Gait Speed Test; Oxford Hip Score; WOMAC; Short Form-12 Health Survey (SF-12)

SUMMARY:
This study aims to explore how well patient self-assessments reflect their actual physical performance following hip replacement surgery. By comparing questionnaire-based scores with practical mobility tests, the study seeks to provide insight into the usefulness of both tools in evaluating recovery after total hip arthroplasty.

DETAILED DESCRIPTION:
Hip replacement surgery is generally effective in reducing pain and restoring movement in patients with hip joint problems. Despite the success of the procedure, some individuals continue to report dissatisfaction due to lingering discomfort or limitations in daily activities. A potential reason for this is the gap between how patients perceive their recovery and their actual physical function.

To better understand this issue, the study evaluates two types of assessment tools. The first group includes patient-reported outcome measures (PROMs), which rely on individuals' personal impressions of their symptoms and abilities. The second group involves physical performance tests that measure mobility and balance under clinical supervision.

Fifty patients who had hip replacement surgery at least six months earlier will take part in the study. Each participant will complete standardized questionnaires and undergo a series of physical tests during one clinic visit. The relationship between the two types of assessments will be analyzed using correlation and regression methods.

This research may help improve follow-up care by identifying whether patient questionnaires alone are sufficient to monitor recovery, or if performance-based tests should also be routinely included in rehabilitation planning.

ELIGIBILITY:
Inclusion Criteria:

* Underwent unilateral primary total hip arthroplasty at least 6 months prior
* Ability to walk independently (with or without assistive device)
* Ability to understand and complete assessments and questionnaires

Exclusion Criteria:

* Revision or bilateral total hip arthroplasty
* Additional lower extremity surgery after the index THA
* Body mass index (BMI) greater than 40 kg/m²
* Neurological, orthopedic, or systemic disorders affecting gait or balance
* Severe cognitive impairment or communication difficulties

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 55 years and older who underwent unilateral primary total hip arthroplasty at least six months prior. All participants were able to walk independently and had sufficient cognitive and communication abilities to complete physical and questionnaire-based assessments.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Correlation Between PROM Scores and Performance-Based Test Results Correlation Between PROM Scores and Performance-Based Test Results Correlation Between PROM Scores and Performance-Based Test Results | Day of assessment (single visit)
  The study will assess the strength and direction of the relationship between patient-reported outcomes (Oxford Hip Score, WOMAC, SF-12) and physical performance test results (Timed Up and Go, Four Square Step Test, 4-Meter Gait Speed Test) using correlation coefficients.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf POLAT, Assoc.Prof., Study Director — Ordu University
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No